CLINICAL TRIAL: NCT06197815
Title: Comparison of Off-site vs. hands-on Assistance for Trainees During ERCP: a Randomized, Controlled, Noninferiority Study
Brief Title: Comparison of Off-site vs. hands-on Assistance for Trainees During ERCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: Department of Endoscopy, Eastern Hepatobiliary Hospital, Second Military Medical University (Unknown); Department of Gastroenterology, The Second Affiliated Hospital Chongqing Medical University (Unknown)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KY20232429
Record Dates: First submitted 2023-12-27; First posted 2024-01-09 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: ERCP Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Off-site assistance group (Experimental): The trainer supervised the trainee's cannulation operation outside the procedure room through a high-definition screen displaying the endoscopic view. Trainees wear headphones, and trainers use intercom to provide the unlimited verbal instructions. The trainer was not allowed into the procedure room and touched the endoscope or accessories until the trainee ask for help or failed to achieve deep biliary cannulation. Then the trainer would then take over and continue with the cannulation. The trainer would halt and correct the trainee's inappropriate maneuvers immediately to avoid unnecessary papillary trauma and potential complications.
  Interventions: Behavioral: The assistance type during ERCP
- Hands-on assistance group (Active Comparator): During trainees' attempted cannulation, the trainer gave unlimited verbal instructions with hands-on assistance limited to only adjustment of scope position if necessary. To avoid unintended cannulation, the trainer was not allowed to touch the control section of the scope or the sphincterotome used for cannulation. However, the trainer would correct any inappropriate maneuvers immediately to avoid unnecessary papillary trauma and potential complications. The trainees could ask for help or stop cannulation at any time if they were not comfortable continuing the procedure. The trainer would then take over and continue with the cannulation.
  Interventions: Behavioral: The assistance type during ERCP

INTERVENTIONS:
Behavioral: The assistance type during ERCP — The senior trainer guides the trainees during ERCP procedure outside the operating room using communication equipment and the screen displaying an endoscopic view.

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is a technically challenging procedure. It takes time to learn the basic skill and at least 180 - 200 cases for trainees to achieve competency in ERCP. Hands-on practice in patients remains the gold standard for ERCP training. It required the trainer to stand by the trainee in the procedure room to assist. There were insufficient patients for most trainees to achieve competence until the trainee graduate. Technology-enabled health care at a distance has profound scientific potential and accordingly has been met with growing interest. We hypothesized that the trainee can be safely guided by a senior trainer off-site with the endoscopic view displayed on a screen. Using the teleguidance, the trainer can even continue to provide guidance when the trainees complete their training and return to their hospitals until they achieve the recommended clinical competency. Given the advantages of the off-site teleguidance, it could be an attractive substitute for hands-on assistance to ERCP training.

The primary aim of this study was to evaluate whether off-site assistance (OA group) could achieve a comparable success rate to standard hands-on assistance (HA group) with regard to the rates of successful selective biliary cannulation during ERCP training.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-90 years who received ERCP
2. Patients with native papilla

Exclusion Criteria:

1. Patients with altered anatomy (Billroth I/II, Roux-en-Y)
2. Type II duodenal stenosis
3. Previously failed cannulation
4. Chronic pancreatitis with stones in the pancreatic head
5. Hemodynamic instability
6. Lactating or pregnant women
7. Inability to give written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 754 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Rates of successful biliary cannulation | 10 minutes
  The percentage of trainee successfully biliary cannulation

SECONDARY OUTCOMES:
Cannulation time | 1 day
Competency score from the trainer and endoscopic video | 1 day
Incidences of PEP and other adverse events | 1 month
Ionizing radiation time | 1 day

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Department of Gastroenterology, The Second Affiliated Hospital Chongqing Medical University, Chongqing, Chongqing Municipality
  - Xijing Hospital of Digestive Diseases, Fourth Military Medical University, Xi'an, Shaanxi
  - Department of Endoscopy, Eastern Hepatobiliary Hospital, Second Military Medical University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No